CLINICAL TRIAL: NCT00002980
Title: A Phase I Study of the Biologic and Clinical Effects of 5-AZA-2'Deoxycytidine (DAC) in Patients With Advanced Malignancies
Brief Title: Decitabine in Treating Patients With Melanoma or Other Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065502; LAC-USC-0C963; NCI-T95-0070
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; primary myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of decitabine in treating patients with stage III or stage IV melanoma or other advanced cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify dosage level(s) of decitabine (DAC) that show biologic activity and acceptable side effects. II. Describe the side effects and toxicity of DAC at the doses studied. III. Determine the steady state DAC serum levels at the doses studied. IV. Document any clinical responses to DAC.

OUTLINE: A dose escalation schedule for the administration of decitabine (DAC) is being used to determine the MTD and biologically active dose. Patients are given two 12 hour continuous infusions per day, for 3 days at each dose level. A minimum of 3 patients are enrolled at each dose level until dose limiting toxicity (DLT) or biologic activity is observed. If DLT or biologic activity is observed at a particular dose level, an additional 3 patients are enrolled, for a total of 6. If 2 or more patients experience DLT, dose escalation is ceased.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Stage III (nonresectable) and IV melanoma, or any other advanced metastatic malignancy for which all standard therapy has failed Must have at least two cutaneous, mucosal or lymph nodal lesions that can be biopsied or one lesion large enough to be biopsied twice

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Hemoglobin at least 9.0 g/dL Platelet count at least 100,000/mm3 WBC at least 3500/mm3 Absolute granulocyte count at least 1500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT less than 2.5 times normal Renal: Creatinine no greater than 1.8 mg/dL Other: Not pregnant Not HIV or hepatitis BsAg positive No major systemic infections No coagulation disorders No major illness of cardiovascular or respiratory systems No symptomatic CNS disease or evidence of cerebral edema

PRIOR CONCURRENT THERAPY: No therapy for cancer within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-05

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (4):
- United States (4):
  - Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Los Angeles County-University of Southern California Medical Center, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California